CLINICAL TRIAL: NCT05713279
Title: Preliminary Clinical Study of Efficacy and Safety of Flunotinib Maleate Tablets Combined With Antiviral Therapy in Patients With Severe Novel Coronavirus (COVID-19) Infection
Brief Title: Study of Flonoltinib Maleate Tablets in the Treatment of Severe Novel Coronavirus (COVID-19) Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZLFM-003-2.0
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FM+SOC (Experimental)
  Interventions: Drug: SOC
- FM安慰剂 +SOC (Placebo Comparator)
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: SOC — In this study, the standard treatment plan (SOC) for COVID-19 in the Department of Respiratory and Critical Care Medicine was used as the best accessible treatment, and the treatment plan principle was based on the latest national guidance document ("Expert Recommendations for Clinical Treatment of Severe Novel Coronavirus Infection Caused by Omicron Variant"; "Diagnosis and Treatment Plan for Novel Coronavirus Infection (Trial Version 10)"; "Diagnosis and Treatment Plan for Severe Cases of Novel Coronavirus Infection (Trial Fourth Edition)"). In this study, the drug flunotinib maleate (FM) 100mg is a class of JAK inhibitors of anti-inflammatory therapy of SOC as standard clinical treatment regimen, and will be used in combination with SOC according to the judgment of the investigator.

SUMMARY:
Flonoltinib Maleate as a JAK/FLT3 dual target inhibitor, previous pharmacological experiments showed that the IC50 inhibition of JAK2 kinase was as low as 0.8 nM, while the IC50 inhibition of JAK1, JAK3 and TYK2 kinases was 26 nM, 39 nM and 2 nM, respectively, and the IC50 of FLT3 kinase was 15 nM. It has high inhibitory activity for JAK2 kinase and good selectivity for JAK family.Multiple pharmacodynamic models evaluating the anti-inflammatory effect of Flonoltinib Maleate showed that Flonoltinib Maleate showed better therapeutic effect than the clinical drug Ruxolitinib with lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old, gender is not limited;
2. COVID-19 infection inclusion criteria: hospitalized with coronavirus (COVID-19) within 14 days, samples collected 72 hours before enrollment confirmed by polymerase chain reaction (PCR) test or antigen test (if due to lack of testing supplies, testing capacity and conditions are limited, but indicate a progressive disease with persistent infection with COVID-19), the investigator judged that the condition was aggravated, and any of the following criteria were met as severe COVID-19 patients:

   Respiratory distress, respiratory rate≥ 30 times/min; At rest, oxygen saturation ≤ 93% when inhaling air; Arterial partial pressure of oxygen (PaO2)/oxygen inhalation concentration (FiO2)≤ 300 mmHg; Clinical symptoms are progressively aggravated, lung imaging shows that the lesions within 24~48h have progressed significantly > 50%.

   Adults with any of the following are defined as critically ill with COVID-19: respiratory failure requiring mechanical ventilation; Appearance of shock; Other organ failure requires ICU monitoring; Severe and critical cases of novel coronavirus infection, collectively referred to as "severe cases". Severe cases can also be managed as severe cases if pneumonia caused by novel coronavirus infection does not meet the diagnostic criteria for severe cases: age > 65 years old, incomplete full vaccination, and more serious chronic diseases (including hypertension, diabetes, coronary heart disease, chronic lung disease, malignant tumors, and immunocompromise, etc.)
3. Patients with risk of progression before enrollment: at least one inflammatory index greater than the upper limit of normal (IL-6, CRP, d-dimer, LDH, ferritin≥ULN) within 2 days;
4. willing and/or able to comply with research-related procedures and assessments;
5. Those who can understand and agree to participate in this research and sign the informed consent form;

Exclusion Criteria:

1. Known or suspected allergy to the test drug and its excipients;
2. Are receiving cytotoxic or biological therapy (such as TNF inhibitors, IL-1 inhibitors, IL-6 inhibitors (tocilizumab, adalimumab, etc.), T cell or B cell targeted therapy (rituximab, interferon, etc.), or Janus kinase (JAK) inhibitors, except for this study.
3. Have received convalescent new coronary pneumonia plasma or intravenous human immunoglobulin; have received clearly effective COVID-19 virus neutralizing antibodies;
4. In addition to the new crown infection, there are other serious infections, suspected serious bacteria, fungal viruses, active tuberculosis, NTM, etc.
5. Known positive for HIV antibody, positive test for active hepatitis B virus (HBsAg positive, HBV-DNA positive or ≥1000 copies/mL), anti-HCV antibody or HCV-RNA positive;
6. Have received a live vaccine within 1 week prior to screening, or are expected to be vaccinated during the study period.
7. Severe liver disease (total bilirubin (TBIL) ≥ 3 times the upper limit of normal value, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥5 times the upper limit of normal value);
8. Those with severe renal insufficiency (glomerular filtration rate ≤ 30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis;
9. Blood routine: neutrophil count < 1.0×109/L, lymphocyte count < 0.2×109/L, platelet < 30×109/L, hemoglobin < 60g/L;
10. Patients with malabsorption syndrome, or any other condition that affects gastrointestinal absorption, requiring intravenous nutrition or unable to take oral medications;
11. Invasive respiratory support or advanced life support, such as ECMO, is required.

Patients who have suffered from malignant tumors in the past 5 years and are currently uncontrolled; (13) Patients who participated in other new drugs or medical devices within 1 month before screening and took the investigational drug and used the investigational device; (14) Pregnant or lactating female patients, female patients with fertility and male patients who refuse to use contraception during the trial and within 6 months after the end of the test; (15) having taken a strong CYP3A inhibitor (such as ketoconazole, clarithromycin, itraconazole) or a strong CYP3A4 inducer (rifampicin) within two weeks before the first dose; (16) Patients with congenital coagulation abnormalities, such as patients with a history of multiple thrombosis and bleeding diseases; (17) Alcohol dependence or drug abuse; The researchers believe that patients with rapid disease progression are unlikely to survive for at least 48 hours after screening; or other factors that are not suitable for participation in the trial。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoints | 28 day
  The primary endpoint will assess the proportion of patients who die or require non-invasive ventilation/high-flow oxygen or invasive mechanical ventilation (including extracorporeal membrane oxygenation [ECMO]) at day 28.
Primary efficacy endpoints | 28 day
  Non-invasive ventilation/high-flow oxygen includes ventilatory support without the use of invasive artificial airways (endotracheal tubes or tracheostomy tubes).
Primary efficacy endpoints | 28 day
  High-flow oxygen includes respiratory support through masks, nasal masks, etc.

SECONDARY OUTCOMES:
Secondary efficacy endpoints | 28 day
  Number of days hospitalized and admitted to the ICU (D1-D28);
Secondary efficacy endpoints | 28 day
  If it is separated from oxygen therapy and maintained for 24 hours or without oxygen in the room, SpO2≥93 can be reached and maintained for 24 hours (D1-D28)
Secondary efficacy endpoints | 14 day
  Duration of symptoms associated with COVID-19 infection (D1-D14)
Secondary efficacy endpoints | 28 day
  The proportion and time of the WHO clinical status rating (from 0 (no viral infection) to 10 (death) decreased by two levels
Secondary efficacy endpoints | 28 day
  To improve clinical time
Secondary efficacy endpoints | 28 day
  Rehabilitation time (D1-D28) (Rehabilitation is defined as a patient meeting any of the minimum 3 scores on the NIAID-OS scale (see Appendix) on the first day or time of study initiation: hospitalization, no need for supplemental oxygen - no ongoing medical care is required; not hospitalized, limited mobility, and/or requiring home oxygen; Not hospitalized and with unlimited activities (also applies to normal discharge home)
Secondary efficacy endpoints | 28 day
  Improvement of inflammatory factor levels.
Secondary efficacy endpoints | 28 day
  Nucleic acid negative time (nucleic acid negative is defined as CT value≥35)

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Zenitar Biomedical Technology Co., Ltd, Chengdu, Sichuan, China